CLINICAL TRIAL: NCT00886652
Title: Results of an Aerobic Exercising Program on Respiratory Muscle Strength in Patients With Adolescent Idiopathic Scoliosis: a Randomized, Controlled Trial
Brief Title: An Aerobic Exercising Program on Respiratory Muscle Strength in Patients With Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Osmar Avanzi, Professor Titular, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIS-301/08
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2009-04

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Scoliosis; Muscle Strength; Respiratory function tests; Exercise therapy
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): The patients of the Exercise group were submitted to a four-month physiotherapy protocol, with three weekly sessions of 60 minutes each, accompanied by a physiotherapist, and consisting of warm-up, aerobic exercise on an electric treadmill, and then winding down and relaxation.
  Each patient in this group was therefore submitted to an average of 48 sessions of exercises, always carried out at the same physiotherapy center.
  Interventions: Other: Aerobic exercise program
- 2 (No Intervention): The patients of the control group were not submitted to any type of physical exercises. Like the patients submitted to the protocol, they were evaluated at the beginning, and again after four months.

INTERVENTIONS:
Other: Aerobic exercise program — Three weekly sessions, with an interval of one day between each, lasting 60 minutes each, and divided into three separate stages: - A 10-minute warm-up (stretching and low intensity aerobic exercises such as slow, gradual walking); - 40 minutes of aerobic exercise on an electric treadmill, with the work intensity maintained at a 60% to 80% of the maximum heart rate; - 10 minutes of winding down and relaxation (stretching exercises, low energy expenditure aerobics and relaxation techniques).
  Arms: Exercise

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) can change the respiratory dynamics and performance of the inspiratory and expiratory muscles, affecting ventilatory capacity. This was a randomized, controlled, open study to test the impact of a physiotherapeutic program of aerobic exercises on respiratory muscle strength, in patients with adolescent idiopathic scoliosis. Patients with AIS were randomly assigned to the aerobic exercise-training program group or the no treatment group. There was a significant increase in Pimax and Pemax in the group which received physiotherapy.

DETAILED DESCRIPTION:
Study Design: This was a randomized, controlled, open study to test the impact of a physiotherapeutic program of aerobic exercises on respiratory muscle strength, in patients with adolescent idiopathic scoliosis (AIS). Objective. To analyze, by means of maximum respiratory pressure measurements, the conditioning of the respiratory muscles after four months of aerobic exercise training. Summary of Background Data. AIS can change the respiratory dynamics and performance of the inspiratory and expiratory muscles, affecting ventilatory capacity.

Methods: Patients with AIS, aged between 10 and 20 years, were randomly assigned to the aerobic exercise-training program group or the no treatment group. They were evaluated for respiratory muscle strength before and after the treatment period, by means of a manometer, and radiographs of the chest and spine. The physical therapy exercise protocol consisted of three weekly sessions, including stretching, aerobic exercises (first mild and then accelerated) and relaxation techniques, for a period of four months.

ELIGIBILITY:
Inclusion Criteria:

* aged between 10 and 20 years
* diagnosed as having adolescent idiopathic scoliosis with a spinal angle of scoliotic deformity of at least 45º, and candidates for surgical correction
* sedentary

Exclusion Criteria:

* spinal angle deformities of less than 45º
* previous operation for spinal correction
* comorbidities (lung, heart or neurological diseases) that could interfere with the understanding of the procedures of this study (both diagnostic and interventional)
* regular physical activity

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Maximum respiratory pressure measurements by means of a manometer: maximum inspiratory pressure (Pimax) and maximum expiratory pressure (Pemax) | Before the start of the proposed exercises, and one day after the last session of the exercise protocol, all the patients were evaluated using a manovacuometer.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Lúcia S Alves, PhD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo; Osmar Avanzi, PhD, Study Chair — Irmandade da Santa Casa de Misericórdia de São Paulo
Locations (1):
- Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Windisch W, Hennings E, Sorichter S, Hamm H, Criee CP. Peak or plateau maximal inspiratory mouth pressure: which is best? Eur Respir J. 2004 May;23(5):708-13. doi: 10.1183/09031936.04.00136104. PMID 15176684
- [Background] Wagener JS, Hibbert ME, Landau LI. Maximal respiratory pressures in children. Am Rev Respir Dis. 1984 May;129(5):873-5. doi: 10.1164/arrd.1984.129.5.873. PMID 6721285
- [Background] Shneerson JM. Cardiac and respiratory responses to exercise in adolescent idiopathic scoliosis. Thorax. 1980 May;35(5):347-50. doi: 10.1136/thx.35.5.347. PMID 7434284
- [Background] dos Santos Alves VL, Stirbulov R, Avanzi O. Impact of a physical rehabilitation program on the respiratory function of adolescents with idiopathic scoliosis. Chest. 2006 Aug;130(2):500-5. doi: 10.1378/chest.130.2.500. PMID 16899851
- [Background] Covey MK, Larson JL, Wirtz S. Reliability of submaximal exercise tests in patients with COPD. Chronic obstructive pulmonary disease. Med Sci Sports Exerc. 1999 Sep;31(9):1257-64. doi: 10.1097/00005768-199909000-00005. PMID 10487366